CLINICAL TRIAL: NCT05487287
Title: Computational Assessment of Hand Motor Skills in Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Hospital Universitario La Paz (Other); Universidad Politecnica de Madrid (Other)
Responsible Party: Sponsor
Other Study IDs: PI-4776
Record Dates: First submitted 2022-06-10; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-05

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ischemic stroke patients with functional deficit of the hand
  Interventions: Device: Kinematic computational analysis of the hand (Leap Motion device)
- Healthy subjects
  Interventions: Device: Kinematic computational analysis of the hand (Leap Motion device)

INTERVENTIONS:
Device: Kinematic computational analysis of the hand (Leap Motion device) — Kinematic computational analysis exercises:
  1. Finger extension
  2. Wrist extension
  3. Finger separation
  4. Finger clamp

SUMMARY:
This is a two phase prospective observational study that aims to validate the use of a motion capture software (Leap Motion) to measure and quantify functional deficits of the hand in stroke patients using a standard battery of exercises. The objectives of this study are:

1. To compare the differences between results of hand kinematic computational analysis in patients with ischemic stroke and healthy subjects.
2. To analyze the relation between hand kinematic computational analysis and clinical scales usually performed to evalutate neurologic deficits in stroke patients.
3. To analyze the relation between hand kinematic computational analysis and stroke lesion on brain MRI.
4. To analyze changes between results of hand kinematic computational analysis in the acute phase of stroke and at three months, and its relation with evolution of neurological evaluation clinical scales, functional clinical scales and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients: clinically stable, with hand functional deficit at the momment they consent to participate in the study. Signed consent to participate.
* Healthy subjects: similar age to stroke patients, without previous clinical history of stroke or any disease that could affect hand motor skills. Signed consent to participate.

Exclusion Criteria:

* Aphasia or cognitive impairment, confusional syndrome or other conditions that could prevent comprehension and acomplishment of the task.
* Plegia or severe paresis of the hand that could prevent adecuate performance of the task.
* Previous stroke.
* Previous dependance.
* Previous diagnosis of any other neurologic disease or condition that could affect hand motricity.
* Life expectancy below three months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cases: 100 subjects with ischemic stroke with functional motor hand deficit Healthy subjects: 100 subjects matched by age with ischemic stroke patients.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Hand kinematic computational analysis | First month
  o compare the differences between results of hand kinematic computational analysis in patients with ischemic stroke and healthy subjects.
Relation between hand kinematic computational analysis and clinical scales | First month
  To analyze the relation between hand kinematic computational analysis and clinical scales usually performed to evalutate neurologic deficits in stroke patients.
Relation between hand kinematic computational analysis and stroke lesion on brain MRI. | First month
  To analyze the relation between hand kinematic computational analysis and stroke lesion on brain MRI.
Results of hand kinematic computational analysis in the acute phase of stroke and at three months, and its relation with evolution of neurological evaluation clinical scales, functional clinical scales and quality of life. | 1 month and three months
  Changes between results of hand kinematic computational analysis in the acute phase of stroke and at three months, and its relation with evolution of neurological evaluation clinical scales, functional clinical scales and quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain